CLINICAL TRIAL: NCT04544397
Title: Outcomes of Second Generation Laser Balloon Ablation for Atrial Fibrillation Assessed by Continuous Rhythm Monitoring
Brief Title: Outcomes of Second Generation Laser Balloon Ablation for Atrial Fibrillation
Acronym: LIGHT-AF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Luigi Sacco University Hospital (Other)
Responsible Party: Principal Investigator, Giovanni B Forleo, Section Head Electrophysiology, Luigi Sacco University Hospital
Other Study IDs: LIGHT-AF
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation Paroxysmal; Atrial Fibrillation, Persistent
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Catheter Ablation for AF — Pulmonary vein isolation (PVI) is the mainstay goal of atrial fibrillation (AF) ablation procedures, especially in paroxysmal AF (PAF), and is recommended during all AF ablation procedures. PVI can be obtained with different techniques, using 3D-mapping systems guiding point-by-point radiofrequency (RF) ablation procedures or balloon-based ablation systems (cryo- or laser balloon), introduced to simplify catheter ablation for AF. In particular, the 2nd generation of visually guided laser balloon ablation system (LB2) makes use of laser energy to achieve PVI, leading to better PV occlusion and isolation compared to the 1st generation.

SUMMARY:
The purpose of this study is to collect data on laser ballon (2nd gen) systems for catheter ablation for AF, in order to determine the safety and the efficacy of this technique.

Moreover, the investigators aim to determine the short and long term outcomes of pulmonary vein isolation evaluating arrhythmia recurrence, especially using continuous rhythm monitoring with implantable loop recorders (ILR).

DETAILED DESCRIPTION:
LIGHT-AF is an observational, multicentric study designed to collect pre-procedural, procedural and follow-up data of consecutive patients that underwent catheter ablation for AF with laser ballon (2nd gen system). A number of 3 enrolling centers is estimated with an overall number of about 100 patients. A minimal follow-up of 3 months is required before analyzing clinical outcomes. The data analysis will focus on implant outcomes and early, mid and long-term recurrence of AF, evaluated with intracardiac rhythm monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Patients with paroxysmal, persistent or long-standing persistent AF
* Patients able to provide written informed consent or have informed consent as provided by a legal representative

Exclusion Criteria:

* Age < 18 years
* Patients unable or unwilling to receive oral anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >/= 18 years, with paroxysmal or persistent AF, that met the indications provided by international guidelines to undergo catheter ablation for AF as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
AF recurrences | 2 years
  Time to first recurrence of symptomatic or asymptomatic atrial tachyarrhythmias

SECONDARY OUTCOMES:
Arrhythmia burden | 2 years
  Percentage of overall time in AF
Redo ablation procedures | 2 years
  Patients requiring a redo ablation procedure, after the first one
Adverse events | 2 years
  Procedural mortality or other adverse events related to the procedure

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS Policlinico San Donato, San Donato Milanese, Milano
  - Ospedale Luigi Sacco - Polo Universitario, Milan, Mi
  - Ospedale San Gerardo - ASST Monza, Monza

IPD SHARING:
Plan to Share IPD: Undecided